CLINICAL TRIAL: NCT04529109
Title: Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6395
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects that are habitual soft contact lens wearers and current wearers of circle/cosmetic contact lenses will be randomized into lens wear sequence (Test/Control).
  Interventions: Device: etafilcon A investigational cosmetic lens 1; Device: etafilcon A investigational cosmetic lens 2
- Control/Test (Experimental): Eligible subjects that are habitual soft contact lens wearers and current wearers of circle/cosmetic contact lenses will be randomized into lens wear sequence (Control/Test).
  Interventions: Device: etafilcon A investigational cosmetic lens 1; Device: etafilcon A investigational cosmetic lens 2

INTERVENTIONS:
Device: etafilcon A investigational cosmetic lens 1 — TEST
Device: etafilcon A investigational cosmetic lens 2 — CONTROL

SUMMARY:
This will be a randomized, double-masked, bilateral, cross-over, 2 treatment by 2 period dispensing study. There will be 4 visits. There will be a 2 to 5 day washout period between treatments.

ELIGIBILITY:
Inclusion Criteria:

-Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
2. Females between 18 and 29 (inclusive) years of age at the time of screening
3. Appear able and willing to adhere to the instructions set forth in this clinical protocol (i.e. willing to wear only the study lenses and not use habitual lenses during the dispensing periods)
4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report
5. Be a current wearer of cosmetic/circle lenses in the last 6 months, by self-report.
6. The subject must be willing to be photographed and/or video-taped
7. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye
8. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye
9. Have spherical best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating
2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg, rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion)
3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion)
4. Any previous or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.).
5. Any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear (at the investigators discretion).
6. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
7. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician)
8. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion)
9. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Frazier Vision, Inc, Tyler, Texas
- Hong Kong (2):
  - Vital Eyecare Center, Mong Kok, Kowloon
  - Sight Enhancement Center, Yau Ma Tei, Kowloon

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 58 subjects were enrolled into this study. Of those enrolled, 56 were dispensed at least 1 study lens, while 2 subjects failed to meet all eligibility criteria. Of those dispensed, 55 subjects completed the study while 1 subject was discontinued.
Groups:
- Test/Control: Subjects randomized to receive the Test lens during the first period and then receive the Control lens during the second period. Note: Washout period between periods 1 and 2 is considered period 1.
- Control/Test: Subjects randomized to receive the Control lens during the first period and then received the Test lens during the second period. Note: Washout period between periods 1 and 2 is considered period 1.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 27 | 29
Completed | 27 | 28
Not Completed | 0 | 1
Not completed — Unsatisfactory Lens Fitting due to Test Article | 0 | 1
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: All subjects who were dispensed a study lens.
Arm/Group | Total
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 41
  American Indian or Alaska Native | 1
  Black or African American | 4
  White | 9
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
  China | 39

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Distance Monocular Visual Acuity (logMAR) Lower Than 0.176 logMAR
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters) under high luminance high contrast lighting condition using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. However, the data was dichotomized as Y=1 if logMAR visual acuity was less than 0.176 logMAR; and Y=0 otherwise. A value of 0.176 logMAR ≅20/30 Snellen Visual Acuity. The proportion of eyes with visual acuity lower than 0.176 logMAR was reported.
Time Frame: 5- Minutes Post-Lens Fitting
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: Eyes
Groups:
- Test (Etafilcon A With Cosmetic Pattern): Subjects that wore the Test lens in either the first or second period of the study.
- Control (Etafilcon A With Cosmetic Pattern): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test (Etafilcon A With Cosmetic Pattern) | Control (Etafilcon A With Cosmetic Pattern)
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 102 | 102
proportion of eyes | 0.9998 | 0.9998
Statistical Analysis 1: Comparison: Test (Etafilcon A With Cosmetic Pattern); Test type: Superiority — The superiority of the Test lens was concluded if the lower limit of the 95% credible interval was above 0.90; Bayesian Binary model; Mean Proportion = 0.9998, 95% CI 2-sided [0.999 to 1.000], Standard Deviation 0.0005 — Interval presented is a 95% Credible interval

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 weeks per subject.
Arm/Group | Test (Etafilcon A With Cosmetic Pattern) | Control (Etafilcon A With Cosmetic Pattern)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04529109/Prot_SAP_000.pdf